CLINICAL TRIAL: NCT06961981
Title: Feasibility, Acceptability, and Preliminary Efficacy of a Remote Vinyasa Yoga Program for Heart Health
Brief Title: Remote Vinyasa Yoga Program for Heart Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Bethany Barone Gibbs, PhD, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2410052950
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-04

CONDITIONS: Hypertension; Cardiovascular Diseases
Keywords: Yoga; vinyasa yoga
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vinyasa Yoga (Experimental): Participants will complete a 12-week, remotely-delivered intervention with three 60-minute vinyasa yoga sessions per week via Zoom, following an adapted Journey into Power yoga sequence by Baron Baptiste. The sessions will incorporate three mind-body components of yoga: through physical yoga poses, mindfulness, and breathing.
  Interventions: Behavioral: Vinyasa Yoga
- Standard Routine (No Intervention): Standard usual routine for 12 weeks

INTERVENTIONS:
Behavioral: Vinyasa Yoga — Each yoga session will begin with 2 minutes of integration poses (Child's Pose, Downward Facing Dog, Ragdoll, and Mountain Pose), followed by ~20 minutes of Sun Salutations A and B (up to 5 of each). The Standing Series, lasting ~25 minutes, will include various standing and balancing poses from the Journey into Power sequence. Seated and supine stretches (including seated stretches, a yoga inversion, a reclined twist) will last ~8 minutes, and the session will conclude with 5 minutes of Savasana for final relaxation.
  Other Names: Flow Yoga
  Arms: Vinyasa Yoga

SUMMARY:
The purpose of this study is to test a 12-week vinyasa yoga (flow yoga) intervention via Zoom. This program will be for 30 individuals with high blood pressure. 15 will receive the intervention and 15 will follow their usual routine. The investigators will determine if this vinyasa yoga program is feasible and acceptable in this population. Investigators will measure and compare blood pressure and other health responses such as physical health and well-being before and after participants complete the intervention or usual care period. The investigators hope to demonstrate that vinyasa yoga is a good option to improve heart health in people with high blood pressure.

Primary Objective - Examine the feasibility, acceptability, and preliminary efficacy of a 12-wk remotely-delivered vinyasa yoga intervention (3 x per week) on cardiovascular (CV) health in adults with hypertension (HTN).

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a resting systolic BP >130 mmHg

Exclusion Criteria:

* Report currently meeting aerobic activity guidelines (150 min/wk)
* Practice yoga regularly (1 or more day/wk in the past month)
* Have physical limitations or a major medical condition contraindicating yoga or assessments
* Have uncontrolled HTN (systolic BP 160 mmHg or diastolic BP 100 mmHg)
* Are currently pregnant or planning to become pregnant within 6 months
* Are not on a stable dose of medications that could affect study outcomes
* Are concurrently enrolled in another lifestyle program
* No vulnerable populations will be included

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Carotid-Femoral Pulse Wave Velocity | Baseline to 12 weeks
  Change from baseline to 12 weeks. Measure of central arterial stiffness (meters/second) measured by oscilometiric pulse wave velocity. A value of 10 m/s and above is classified as an unfavorable value.

SECONDARY OUTCOMES:
Change in systolic blood pressure | Baseline to 12 weeks
  Change from baseline to 12 weeks. Measure of pressure in the arteries when the heart beats (millimeters of mercury) measured by an automated blood pressure device with an oscillometric cuff. A value of less than 120 mmHg is considered normal, elevated is a value 120-129 mmHg, and high blood pressure is any value 130 or above.
Change in diastolic blood pressure | Baseline to 12 weeks
  Change from baseline to 12 weeks. Measure of pressure in the arteries between heart beats (millimeters of mercury) measured by an automated blood pressure device with an oscillometric cuff. A value of less than 80 mmHg is considered normal, and high blood pressure is any value 80 or above.
Change in augmentation pressure | Baseline to 12 weeks
  Change from baseline to 12 weeks. Difference in pressure (millimeters of mercury) measured by oscilometiric pulse wave analysis. A value between 20 and 80 mmHg is considered within the normal range, while values at or above 80 mmHg are regarded as unfavorable and may indicate increased cardiovascular risk.
Change in augmentation index | Baseline to 12 weeks
  Change from baseline to 12 weeks. Measure of systemic arterial stiffness (%), measured by oscillometric pulse wave analysis. A value under 33% is considered normal while a value above 33% is considered unfavorable.
Change in mean heart rate | Baseline to 12 weeks
  Change from Baseline to 12 weeks. Measure of the number of heart beats in a minute (beats per minute) measured by a heart rate sensor. A value below 100 is considered normal while values above 100 are unfavorable.
Change in standard deviation of normal R-R Intervals | Baseline to 12 weeks
  Change from Baseline to 12 weeks. A measure of heart rate variability measuring overall variation between R-R intervals (milliseconds) measured by a heart rate sensor recording R-R intervals. Typically, a higher value is considered better for this outcome while a lower value is considered unfavorable.
Change in root mean square of successive differences | Baseline to 12 weeks
  Change from Baseline to 12 weeks. A measure of heart rate variability measuring variability and parasympathetic activity (milliseconds) measured by a heart rate sensor recording R-R intervals. Typically, a higher value is considered better for this outcome while a lower value is considered unfavorable.
Change in high frequency heart rate variability | Baseline to 12 weeks
  Change from Baseline to 12 weeks. A measure of heart rate variability measuring parasympathetic nervous system activity (milliseconds squared) measured by a heart rate sensor recording R-R intervals. Typically, a higher value is considered better for this outcome while a lower value is considered unfavorable.
Change in low frequency heart rate variability | Baseline to 12 weeks
  Change from Baseline to 12 weeks. A measure of heart rate variability measuring sympathetic nervous system activity (milliseconds squared) measured by a heart rate sensor recording R-R intervals. Typically, a lower value is considered better for this outcome while a higher value is considered unfavorable.
Change in low frequency to high frequency ratio | Baseline to 12 weeks
  Change from Baseline to 12 weeks. A measure of heart rate variability measuring the ratio of sympathetic and parasympathetic nervous system activity (unitless) measured by a heart rate sensor recording R-R intervals. Typically, a lower value is considered better for this outcome while a higher value is considered unfavorable.
Change in body mass index | Baseline to 12 weeks
  Change from Baseline to 12 weeks. A measure of body fat based on height and weight (kilograms per meters squared) measured by height (stadiometer) and weight (scale). An individual is considered underweight if their BMI is <18.5 kg/m2, normal weight if their BMI ranges from 18.5 to 24.9 kg/m2, overweight if their BMI ranges from 25-29.9 kg/m2, and obese if their BMI is 30.0 kg/m2 or above.
Change in waist-to-hip-ratio | Baseline to 12 weeks
  Change from Baseline to 12 weeks. Measure of the ratio of the circumference of the waist and hip (unitless) measured by a flexible tape measure. For females, a value of <0.85 is ideal with values above this threshold being unfavorable. For males, a value of <0.90 is ideal with values above this threshold being unfavorable.
Change in total body fat percentage | Baseline to 12 weeks
  Change from Baseline to 12 weeks. Estimate of body fat as a percent of total body weight (percent) measured by bioelectrical impedance analysis. Generally, for females, a value of 8-30% would be considered acceptable, and above 30% is considered unfavorable (overweight or obese). Generally, for males, a value of 5-20% would be considered acceptable, and above 20% is considered unfavorable (overweight or obese).
Change in fat mass | Baseline to 12 weeks
  Change from Baseline to 12 weeks. Estimate of fat mass in the body (pounds) measured by bioelectrical impedance analysis. Higher values suggest higher fat mass in the body (typically an unfavorable finding) while lower values are suggestive of lower fat mass in the body (typically a favorable finding).
Change in fat free mass | Baseline to 12 weeks
  Change from Baseline to 12 weeks. Estimate of non-fat mass in the body (pounds) measured by bioelectrical impedance analysis. Typically, higher values indicate more fat free mass (favorable) and lower values indicate less fat free mass (unfavorable).
Change in skeletal muscle mass | Baseline to 12 weeks
  Change from Baseline to 12 weeks. Estimated weight of skeletal muscle in the body (pounds) measured by bioelectrical impedance analysis. Typically, a higher value indicates more skeletal muscle mass (favorable) while a lower value indicates less skeletal muscle mass (unfavorable).
Change in estimated maximal oxygen consumption (VO2) | Baseline to 12 weeks
  Change from Baseline to 12 weeks. Difference in estimated maximal oxygen uptake (mL/kg/min), reflecting changes in cardiovascular fitness. Estimated maximum oxygen uptake (milliliters of oxygen per kilogram of body weight per minute) derived from a submaximal modified Balke treadmill test. Higher values are better for this measurement. Poorer outcomes vary for females and males and by age groups. Females VO2 Max that is considered poor: 18-29 yrs= <34 mL·kg-¹·min-¹, 30-39 yrs= <26 mL·kg-¹·min-¹, 40-49 yrs= <23 mL·kg-¹·min-¹, 50-59 yrs= <21 mL·kg-¹·min-¹, 60-65 yrs= <18 mL·kg-¹·min-¹. Males VO2 Max that is considered poor: 18-29 yrs= <43 mL·kg-¹·min-¹, 30-39 yrs= <37 mL·kg-¹·min-¹, 40-49 yrs= <32 mL·kg-¹·min-¹, 50-59 yrs= <25 mL·kg-¹·min-¹, 60-65 yrs= <22 mL·kg-¹·min-¹.
Change in 1-repetition maximum testing - Seated chest press | Baseline to 12 weeks
  Change from Baseline to 12 weeks. A measure of muscular strength (in pounds), determined through a 1-repition maximum test using a seated chest press machine. A higher weight indicates higher muscular strength.
Change in 1-repetition maximum testing - Seated leg press | Baseline to 12 weeks
  Change from Baseline to 12 weeks. A measure of muscular strength (in pounds), determined through a 1-repition maximum test using a seated leg press machine. A higher weight indicates higher muscular strength.
Change in time-based muscular endurance tests - wall sit | Baseline to 12 weeks
  Change from Baseline to 12 weeks. Duration of maintaining a position (seconds) measured by performing a wall sit. A longer duration would indicate better muscular endurance.
Change in Time-based muscular endurance test - plank | Baseline to 12 weeks
  Change from Baseline to 12 weeks. Duration of maintaining a position (seconds) measured by performing a plank hold. A longer duration maintaining good form in a plank position would indicate better muscular endurance.
Change in count-based muscular endurance test - push-up test | Baseline to 12 weeks
  Change from Baseline to 12 weeks. Maximum number of repetitions of push-ups performed in one session (count), measured by performing push-ups until fatigue. A higher count would indicate better muscular endurance.
Change in upper body flexibility | Baseline to 12 weeks
  Change from Baseline to 12 weeks. Shoulder and hamstring/low back flexibility (centimeters), measured by a back scratch and sit-and-reach test. A positive value would indicate better upper body flexibility, while a negative value would indicate worse upper body flexibility.
Change in lower body flexibility | Baseline to 12 weeks
  Change from Baseline to 12 weeks. Hamstring and low back flexibility (centimeters), measured by a sit-and-reach test. Higher values indicate better lower body flexibility.
Change in perceived stress | Baseline to 12 weeks
  Change from Baseline to 12 weeks. A score is determined from responses to the Perceived Stress Scale survey. Scores range from 0 to 40, with 0-13 typically indicating low stress, 14-26 moderate stress, and 27-40 high stress.
Change in perceived depressive symptoms | Baseline to 12 weeks
  Change from Baseline to 12 weeks. A score is determined from responses to the Center for Epidemiological Studies Depression Scale-Short Form. Scores range from 0-20 with higher values indicating greater depressive symptoms.
Change in perceived sleep | Baseline to 12 weeks
  Change from Baseline to 12 weeks. A global score is determined from responses to the Pittsburgh Sleep Quality Index Questionnaire. Scores range from 0 to 21 with a score of 5 or higher suggestive of sleep difficulties.
Change in body image perception | Baseline to 12 weeks
  Change from Baseline to 12 weeks. A score is determined from responses to the Body Self-Image Questionnaire Short Form. Scores can range from 27 to 135 with higher scores suggesting more body image dissatisfaction.
Change in perceived anxiety symptoms | Baseline to 12 weeks
  Change from Baseline to 12 weeks. A score is determined from responses to the Generalized Anixety Disorder-7 survey. Scores range from 0 to 21 with higher values represting more anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Barone Gibbs, PhD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States